CLINICAL TRIAL: NCT03865511
Title: MELROSE: Phase 2 Study Evaluating MEchanisms of Resistance on Tumor Tissue and Liquid Biopsy in Patients With EGFR Mutated Nonpretreated Advanced Lung Cancer Receiving OSimErtinib Until and Beyond Radiological Progression : the MELROSE Trial
Brief Title: MEchanisms of Resistance in EGFR Mutated Nonpretreated Advanced Lung Cancer Receiving OSimErtib
Acronym: MELROSE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC18_0287
Record Dates: First submitted 2019-02-27; First posted 2019-03-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAGRISSO® 80mg (Osimertinib) (Experimental): Oral administration of TAGRISSO® 80mg (Osimertinib) as a single daily dose until disease progression or unacceptable toxicity.
  Tumor biopsies performed at baseline and clinical progression. ctDNA analysis by Collection of plasma (two 10-ml Streck tubes) at each time point indicated in the trial.
  Interventions: Drug: TAGRISSO® 80mg (Osimertinib); Genetic: Tumor biopsies; Genetic: ctDNA analysis

INTERVENTIONS:
Drug: TAGRISSO® 80mg (Osimertinib) — Oral administration of TAGRISSO® 80mg (Osimertinib) as a single daily dose until disease progression or unacceptable toxicity.
Genetic: Tumor biopsies — Tumor biopsies performed at baseline and clinical progression will be processed (fixed) on site, and sent to Nantes University Hospital for analysis.
  The following analysis will be performed:
  1. Analyses performed on a regular basis, in order to allow subsequent inclusion in other clinical trials :
     * C797S testing (digital PCR)
     * MET amplification (dPCR/FISH)
     * Histological examination of the tissue sample (to identify small cell transformation)
     * Expression of proteins by immunohistochemistry: PD-L1 (Ventana SP263 antibody); CD73 ; CD4; CD8.
  2. At the end of inclusions, deep sequencing analysis to identify acquired mutations and copy number variations (amplifications).
Genetic: ctDNA analysis — ctDNA analysis by Collection of plasma (two 10-ml Streck tubes) at each time point indicated in the trial.
  These samples will be sent at room temperature by courier to the central laboratory (Nantes University Hospital). There they will be centrifuged, and plasma will be frozen (-80°C).
  Analyses :
  * Detection of the EGFR activating mutation in plasma at baseline By dPCR (characterization of patients enrolled)
  * Detection of the EGFR activating mutation at d7 and m1 by dPCR (early detection of response to osimertinib)
  * Analysis of the plasma samples collected at clinical progression in order to identify acquired mechanisms of resistance by NGS (and comparison with analysis of the biopsies).
  * Kinetics studies of the alterations

SUMMARY:
Osimertinib is an epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKI) that is selective for both EGFR-TKI sensitizing and T790M resistance mutations in patients with non-small-cell lung cancer.

The AURA 3 study (T790M-positive advanced non-small-cell lung cancer in progression after first-line EGFR-TKI therapy, shown that the median duration of progression-free survival was significantly longer with osimertinib than with platinum therapy plus pemetrexed (10.1 months vs. 4.4 months p<0.001).

In addition, clinical data show that patients with mutated EGFR NSCLC receiving osimertinib in first line, presented an objective response rate of 77 % with a disease control rate of 98 % and a median PFS was 19.3 months.

Finally, The FLAURA study randomized phase 3 study clearly demonstrated the superiority of osimertinib compared with erlotinib or gefitinib in EGFR mutated nonpretreated NSCLC (median PFS of 18.9 months versus 10.2 months).

However, several issues remain unknown or debated :

* What are the mechanisms of resistance to osimertinib prescribed in first-line?
* What are the consequences of prolonged exposure to osimertinib on the expression of markers of response to immunotherapy?
* Is there an association between kinetic parameters of ctDNA (circulating tumor DNA) and prediction of response to osimertinib and/ or and prediction of therapeutic escape under osimertinib? In order to respond to all these questions, this phase II trial will be the first to systemically analyze the mechanisms of resistance to Osimertinib based on the analysis of biopsy, and collection of plasma from all patients during the course of treatment.

ELIGIBILITY:
Inclusion Criteria :

1. Male or female, aged at least 18 years.
2. Informed consent signed prior to any study speciﬁc procedures, sampling, and analyses.
3. Pathologically conﬁrmed adenocarcinoma of the lung (e.g., this may occur as systemic recurrence after prior surgery for early stage disease or patients may be newly diagnosed with Stage lIIB/ IV disease). Patients with mixed histology are eligible if adenocarcinoma is the predominant histology.
4. Locally advanced or metastatic NSCLC (Non-small-cell lung carcinoma), not amenable to curative surgery or radiotherapy.
5. The tumour harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19 deletions, L858R), either alone or in combination with other EGFR mutations.
6. Patients must be treatment-naive for advanced NSCLC and eligible to receive ﬁrst-line treatment with osimertinib
7. Subjects affiliated to an appropriate health insurance
8. World Health Organization Performance Status of 0 to 1 with no clinically signiﬁcant deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
9. At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline as 10 mm in the longest diameter (except lymph nodes which must have a short axis of 15 mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), and which is suitable for accurate repeated measurements.
10. Female patients should be using adequate contraceptive measures, should not be breast feeding, and must have a negative pregnancy test prior to ﬁrst dose of study drug; or female patients must have an evidence of non-child-bearing potential by fulﬁlling one of the following criteria at screening:

    * Post-menopausal deﬁned as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
    * Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution.
    * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.
11. Male patients should be willing to use barrier contraception, i.e., condoms

Exclusion Criteria :

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
2. Previous enrolment in the present study
3. Treatment with any of the following:

   * Prior treatment with any systemic anti-cancer therapy for advanced NSCLC including standard chemotherapy, biologic therapy, immunotherapy, or any investigational drug.
   * Prior treatment with an EGFR-TKI. including osimertinib
   * Major surgery (excluding placement of vascular access) within 4 weeks of the ﬁrst dose of study drug.
   * Radiotherapy treatment to more than 30% of the bone marrow or with a wide ﬁeld of radiation within 4 weeks of the ﬁrst dose of study drug.
   * Treatment with an investigational drug within ﬁve half-lives of the compound or any of its related material, if known.
4. Any concurrent and/or other active malignancy that has required systemic treatment within 2 years of ﬁrst dose of study drug.
5. Any unresolved toxicities from prior systemic therapy (e. g., adjuvant chemotherapy) greater than CTCAE grade l at the time of starting study drug with the exception of alopecia, prior platinum-therapy related neuropathy grade 2.
6. Spinal cord compression, symptomatic and unstable brain metastases except for those patients who have completed definitive therapy, and have had a stable neurological status for at least 2 weeks after completion of definitive therapy. Patients may be on corticosteroids to control brain metastases if they have been on a stable dose for 2 weeks (14 days) prior to the start of study treatment and are clinically asymptomatic.
7. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol; or active infection including hepatitis B, hepatitis C and human immunodeﬁciency virus (HIV). Screening for chronic conditions is not required.
8. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous signiﬁcant bowel resection that would preclude adequate absorption of osimertinib.
9. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 ECGs, using the screening clinic ECG machine-derived QTc value.
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250 msec.
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events suchas heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in ﬁrst-degree relatives or any concomitant medication known to prolong the QT interval.
   * Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
10. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values.

    * Absolute neutrophil count <1.5 x 109/L.
    * Platelet count <100 x 109/L.
    * Haemoglobin <90 g/L.
    * Alanine aminotransferase (ALT) >2.5x the upper limit of normal (ULN) if no demonstrable liver metastases or >5 x ULN in the presence of liver metastases
    * Aspartate aminotransferase (AST) >2.5 x ULN if no demonstrable liver metastases or >5xULN in the presence of liver metastases.
    * Total bilirubin >1.5 x ULN if no liver metastases or >3 x ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases.
    * Creatinine >1.5 x ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation); conﬁrmation of creatinine clearance is only required when creatinine is >1.5 x ULN.
11. Women who are breast feeding
12. History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib
13. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
14. Adults under a legal protection regime (guardianship, trusteeship, judicial safeguard)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Examination of the genetic profile at the point of disease progression in EGFRm+ (mutated Epidermal Growth Factor Receptor) patients receiving osimertinib as first-line EGFR TKI therapy compared to baseline. | At clinical disease progression (approximately 22 months)
  Analyze of the proportion of patients with a given genetic marker on tumor biopsy (including, but not limited to, EGFR mutations, HER2 (Human Epidermal Growth factor receptor 2), and cMET expression and/or amplification) at the point of clinical disease progression.

SECONDARY OUTCOMES:
Clinical objective : To assess efficacy of Osimertinib | Every 3 months up to one year after first study dose
  Progression free survival rate at one year defined by time from first study dose to first event between Radiological Progression Disease and death, or one year if no event. The rPFS is defined according to RECIST 1.1.
Clinical objective : To assess efficacy of Osimertinib | Every 3 months until radiological disease progression (approximately 22 months)
  Radiological Progression Free Survival (rPFS): Time from first study dose to first event between rPFS or death. The rPFS is defined according to RECIST 1.1.
Clinical objective : To assess efficacy of Osimertinib | Every month until clinical disease progression (approximately 22 months)
  Clinical Progression Free Survival (cPFS): Time from first study dose to off-osimertinib.
Clinical objective : To assess efficacy of Osimertinib | From first dose to end of study or date of death from any cause, whicheever comes first, assessed every 3 months (approximately 48 months)
  Overall survival
Clinical objective : To assess efficacy of Osimertinib | every 3 months until radiological disease progression (approximately 22 months)
  Objective Response Rate (ORR)
Clinical objective : To assess efficacy of Osimertinib: Duration of Response (DoR): Disease Control Rate (DCR) | every 3 months until radiological disease progression (approximately 22 months)
  Duration of Response (DoR): Disease Control Rate (DCR)
Clinical objective : To assess safety of Osimertinib with Monitoring of Adverse events (grade 3 and 4) | monthly from first study dose until 15 days after last study dose
  Monitoring of Adverse events (grade 3 and 4)
Biological objective : To evaluate the consequence of osimertinib treatment on the expression of targets of immune check point inhibitors | At baseline and at clinical disease progression (approximately 22 months)
  By the study of the expression of molecules involved in the efficacy of check point inhibitors determined by immunohistochemistry (PD-L1; CD73; CD4; CD8) on tumor tissue collected at progression
Biological objective : To evaluate diagnostic accuracy of ctDNA to detect mutation | At baseline and monthly until clinical disease progression (approximately 22 months)
  Analyze of mutation at progression on tumor tissue and ctDNA
Biological objective : To observe if the presence of ctDNA at baseline is a prognostic factor of clinical progression disease | At baseline and monthly until clinical disease progression (approximately 22 months)
  Analyze of the presence of tumors ctDNA at baseline, clinical progression disease
Biological objective : To demonstrate that the early kinetics of ctDNA is an indicator of response to osimertinib | At baseline and monthly until clinical disease progression (approximately 22 months)
  Analyze of absolute quantities of ctDNA molecules presenting the EGFR mutation identified in the tumor, clinical progression disease
Biological objective : To measure the biological progression (bPFS) in patients treated with osimertinib | At baseline and monthly until clinical disease progression (approximately 22 months)
  Serial monitoring in ctDNA of molecular alterations identified in tissues collected at progression
Biological objective : To compare the genetic profile of the ctDNA and the tumor biopsy | At baseline and at clinical disease progression (approximately 22 months)
  Analyze of the EGFR mutation identified in the tumor biopsy and in the ctDNA
Biological objective : To compare the kinetic of appearance of EGFR mutation and radiological and clinical progression disease | At baseline and monthly until clinical disease progression (approximately 22 months)
  Analyze of the absolute quantities of ctDNA molecules presenting the EGFR mutation monthly, radiological and clinical progression disease

CONTACTS AND LOCATIONS:
Overall Officials: Jaafar BENNOUNA, MD,PhD, Principal Investigator — Nantes University Hospital
Locations (17):
- France (17):
  - CHU d'ANGERS, Angers
  - Crlcc Francois Baclesse, Caen
  - CH de Cholet, Cholet
  - C H I Créteil, Créteil
  - CHD Vendée, La Roche-sur-Yon
  - Chu Grenoble, La Tronche
  - CH Le Mans, Le Mans
  - Hôpital Calmette CHRU de Lille, Lille
  - AP-HM Hôpital Nord Marseille, Marseille
  - CH DU MOENCHSBERG - Hôpital Emile Muller, Mulhouse
  - CHU de Nantes, Nantes
  - Institut Curie, Paris
  - AP-HP Hôpital Tenon, Paris
  - Chru Pontchaillou, Rennes
  - Chru Strasbourg, Strasbourg
  - Chits Ch Sainte Musse, Toulon
  - Chu Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bennouna J, Girard N, Audigier-Valette C, le Thuaut A, Gervais R, Masson P, Marcq M, Molinier O, Cortot A, Debieuvre D, Cadranel J, Lena H, Moro-Sibilot D, Chouaid C, Mennecier B, Urban T, Sagan C, Perrier L, Barlesi F, Denis MG. Phase II Study Evaluating the Mechanisms of Resistance on Tumor Tissue and Liquid Biopsy in Patients With EGFR-mutated Non-pretreated Advanced Lung Cancer Receiving Osimertinib Until and Beyond Radiologic Progression: The MELROSE Trial. Clin Lung Cancer. 2020 Jan;21(1):e10-e14. doi: 10.1016/j.cllc.2019.09.007. Epub 2019 Oct 1. PMID 31648999